CLINICAL TRIAL: NCT07403734
Title: Evaluation of the Efficacy of Bilateral Lumbar Erector Spinae Plane Block (ESPB) on Postoperative Analgesia, Early Mobilization, and Length of Hospital Stay in Patients Undergoing Lumbar Disc Herniation Repair Surgery
Brief Title: Evaluation of the Postoperative Efficacy of Bilateral Lumbar Erector Spinae Plane Block (ESPB) in Patients Undergoing Lumbar Disc Herniation Repair Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Muzaffer GENCER, Associate Professor Doctor, Başakşehir Çam & Sakura City Hospital
Other Study IDs: BSH-ANES-MTK-01
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Opioid Consumption, Postoperative; ESPB; Postoperative Pain; Plane Blocks; Lumbar Disc Herniation; Hospital Stay Time; Patient Satisfaction
Keywords: lumbar erector spinae plane block; postoperative pain; espb; lumbar disc hernia repair surgery
MeSH Terms: conditions — Pain, Postoperative; Intervertebral Disc Displacement; Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ESP Block Group: Patients undergoing single-level lumbar disc herniation repair surgery who receive bilateral lumbar erector spinae plane block with 0.25% bupivacaine (20 ml per side, total 40 ml) under ultrasound guidance 30 minutes prior to anesthesia induction, in addition to standardized general anesthesia and postoperative patient-controlled analgesia.
- Control Group (No Block): Patients undergoing single-level lumbar disc herniation repair surgery who receive standardized general anesthesia and postoperative patient-controlled analgesia without erector spinae plane block.

SUMMARY:
This prospective observational study aims to evaluate the efficacy of bilateral lumbar erector spinae plane (ESP) block in providing effective postoperative analgesia and its potential impact on early mobilization and length of hospital stay in patients undergoing surgical repair of lumbar disc herniation.

Regional anesthesia techniques, particularly erector spinae plane blocks, have become an integral component of multimodal analgesia strategies in postoperative pain management. The ESP block has demonstrated effective analgesia across a wide spectrum of thoracic and abdominal surgeries and is increasingly utilized due to its ease of application and safety profile. By implementing multimodal analgesic techniques, this study seeks to achieve effective pain control, reduce opioid consumption and associated complications, facilitate early mobilization, decrease hospital length of stay, and enhance patient comfort.

DETAILED DESCRIPTION:
With the increasing use of ultrasound in recent years and the advantages it brings, the application of regional anesthesia methods such as truncal and peripheral nerve blocks in postoperative pain management has become the most important part of multimodal analgesia strategies. Among regional techniques, the erector spinae plane block has been shown to provide effective analgesia after many types of surgery and is being used increasingly. The erector spinae plane block provides effective analgesia in a wide spectrum of thoracic and abdominal surgeries such as thoracotomy, cholecystectomy, and bariatric surgery, and at the same time, because it is an easy and safe block, it is finding an increasingly expanding place in daily practice in the treatment of chronic and acute pain. The use of multimodal techniques in postoperative analgesia management aims to provide effective analgesia, thereby reducing opioid consumption and related complications, ensuring early mobilization and shorter hospital stay, and increasing patient comfort.

Lumbar disc herniation repair surgery is associated with significant postoperative pain that can negatively impact patient recovery, mobilization, and overall satisfaction. Postoperative pain control has a significant impact on earlier ambulation, better functional recovery, and patient satisfaction. At the same time, optimal pain management is of great importance in contributing to the reduction of the duration of hospital stay and the risk of adverse events.

This study was planned to investigate whether the Erector Spinae Plane Block provides effective postoperative analgesia in patients undergoing lumbar disc herniation repair surgery, and whether it has a positive effect on early mobilization and hospital length of stay. The study aims to demonstrate the effectiveness of the ESP block in reducing postoperative pain, decreasing narcotic analgesic consumption and protecting patients from the side effects of narcotic analgesics, facilitating early mobilization of patients, shortening hospital stay duration, and increasing patient comfort.

Erector spinae plane block (ESPB) was first described by Forero et al. in 2016, with ultrasound-guided local anesthetic injection between the erector spinae muscle and the transverse process of the thoracic vertebra providing effective analgesia for thoracic neuropathic pain. Since then, the ESPB has been widely used for various surgical procedures and has demonstrated consistent efficacy. The mechanism of action involves the spread of local anesthetic to the dorsal and ventral rami of spinal nerves in the interfascial plane, providing extensive dermatomal coverage. For lumbar spine surgery, bilateral lumbar ESPB has shown promise in providing satisfactory postoperative analgesia.

Since the erector spinae plane block is applied to specific anatomical regions defined under ultrasound guidance by a single experienced anesthesiologist (who has performed this block at least 20 times) and the local anesthetic spread is visually monitored, major differences in block effectiveness between patients are not expected. The procedure will be performed with the patient in a sitting position, targeting the area between the L2-4 transverse process and the erector spinae muscle (anterior to the muscle), using 20 mL of 0.25% bupivacaine bilaterally with ultrasound guidance using a convex probe. The application is bilateral and a total of 40 ml of local anesthetic solution will be used. After the procedure, dermatomal mapping will be performed at 30 minutes using a hot-cold test to evaluate block effectiveness in all patients.

Bilateral Lumbar Erector Spinae Plane Block (ESP) or no block (control) will be applied preoperatively to patients hospitalized in the neurosurgery clinic who come to the operating room to undergo single-level lumbar disc herniation repair surgery, after the necessary information is provided and informed consent is obtained. All patients, whether or not they received a block, will receive postoperative intravenous analgesia with patient-controlled analgesia (PCA) devices set with no basal infusion, a lockout time of 30 minutes, a bolus dose of 5 ml, containing tramadol 4 mg/ml. Data will be obtained and recorded from the PCA devices regarding when the patients' first analgesic need arose, the total number of analgesic demands and at what times they occurred, and the total tramadol dose administered.

Pain is a subjective symptom and will be questioned with the Numeric Rating Scale (NRS), a standardized scale, in order to minimize differences between patients. At predetermined time points in the recovery unit at 0, 15th, 30th, and 60th minutes, and during ward follow-up at 2nd, 6th, 12th, and 24th hours, the patients' pain scores with the Numeric Rating Scale (NRS) (0-10; 0-3: mild pain, 4-6: moderate pain, 7-10: severe pain) will be evaluated at rest, with deep breathing, and with coughing. The need for rescue analgesia in the recovery unit (if NRS pain score is 4 or higher out of 10) will be recorded. For postoperative nausea-vomiting evaluation, the Postoperative Nausea Vomiting Impact Scale Score will be used.

In both groups, patients' demographic data, surgical duration, anesthesia duration, intraoperative hemodynamic parameters, the time of first analgesic need if additional analgesic was required along with its content and dose, patient satisfaction scores at postoperative 24 hours (0: not satisfied at all, 5: very satisfied), time to first mobilization, hospital length of stay, and data on complications related to the applied blocks will be recorded and followed. The anesthesiologist who applies the block, the anesthesiologist who follows the patient perioperatively, and the anesthesiologist who performs patient follow-ups and records data at predetermined time points after surgery will be different.

All patients will receive standardized general anesthesia. Premedication with intravenous midazolam 0.03 mg/kg will be administered when patients arrive at the preoperative waiting area. All blocks will be performed in the block room after sedation and monitored with SpO2, electrocardiography, and noninvasive blood pressure (NIBP). After the procedure, the patient will be taken to the operating table and electrocardiography (ECG), temperature, noninvasive blood pressure, and peripheral oxygen saturation (SpO2) will be monitored. For anesthesia induction, all patients will receive midazolam 0.05 mg/kg, fentanyl 1 mcg/kg, propofol 2-3 mg/kg, and rocuronium 0.6 mg/kg. After induction, anesthesia maintenance will be provided with a flow of 2 L/min, 50% oxygen-air mixture, sevoflurane 2%, and remifentanil 0.05 mcg/kg/min. All patients will receive 8 mg ondansetron as a nausea-vomiting protocol routine in our clinic. At the end of the operation, 1 g paracetamol and 1 mg/kg tramadol will be administered and patients will be awakened. To eliminate neuromuscular blockade, 2-3 mg/kg sugammadex will be administered to patients during awakening.

The study will be conducted at Başakşehir Çam and Sakura City Hospital, Department of Neurosurgery, between July 1, 2024 and July 1, 2025. Data collection will span 6 months, followed by 3 months for statistical analysis and 3 months for manuscript preparation, with completion planned in a total of 1 year.

Statistical analysis will be performed using G-Power (Ver. 3.1.9.4) and SPSS 22.0 software. For categorical variables, number and percentage; for quantitative data, minimum, maximum, mean and standard deviation analyses will be performed. Normal distribution analysis of the data will be performed with Kolmogorov-Smirnov and Shapiro-Wilk tests. Parametric tests (t-test, ANOVA, etc.) will be performed for normally distributed data, and non-parametric tests (Mann-Whitney U, Kruskal-Wallis, etc.) will be performed for non-normally distributed data. Correlation test will be performed for relational analysis and regression test will be performed for effect analysis. In all analyses, a p value < 0.05 will be considered significant.

Since there are no additional interventions or medications to be applied to patients beyond routine clinical practice due to the study, no additional risk is expected. The aim is to demonstrate the effectiveness of the Erector Spinae Plane Block in lumbar disc herniation surgery and implement it routinely in our clinic, thereby reducing postoperative pain in patients, reducing narcotic analgesic consumption and protecting them from the side effects of narcotic analgesics, ensuring early mobilization of patients, shortening hospital stay duration, and increasing patient comfort.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* Age 18-70 years
* Patients scheduled to undergo single-level lumbar disc herniation repair surgery
* American Society of Anesthesiologists (ASA) physical status classification I, II, or III
* Willing to participate in the study (voluntary participation)
* Fully oriented and able to cooperate with study procedures

Exclusion Criteria:

* ASA physical status classification > III
* Patients who refuse to participate in the study
* Age < 18 years or > 70 years
* Active infection at the site of block procedure
* Previous lumbar disc herniation surgery
* Chronic pain condition with continuous analgesic use
* Coagulopathy or bleeding disorders
* Patients unable to cooperate with postoperative pain assessments
* Known allergy to local anesthetic agents
* Body Mass Index (BMI) > 35 kg/m²
* Renal insufficiency
* Hepatic insufficiency

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18-70 years with single-level lumbar disc herniation scheduled for surgical repair at Başakşehir Çam and Sakura City Hospital, Department of Neurosurgery. Participants must be ASA I-III, able to provide informed consent, and capable of cooperating with postoperative assessments. Patients with previous lumbar surgery, chronic pain, contraindications to regional anesthesia, or significant comorbidities will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in Postoperative Pain Scores Using Numeric Rating Scale (NRS) | Assessed at 0, 15, 30, 60 minutes in the recovery unit and at 2, 6, 12, and 24 hours postoperatively on the ward (total assessment period: 24 hours)
  Pain intensity will be measured using the 11-point Numeric Rating Scale (NRS: 0-10), where 0 represents "no pain" and 10 represents "worst pain imaginable." Pain scores will be assessed in three conditions: at rest, during deep breathing, and during coughing. The primary analysis will focus on pain scores at rest during the first 24 hours postoperatively.

SECONDARY OUTCOMES:
Total Opioid (Tramadol) Consumption | 24 hours postoperatively
  Total amount of tramadol consumed via patient-controlled analgesia (PCA) device during the postoperative period, measured in milligrams.
Time to First Analgesic Request | From recovery unit arrival (0 minutes) up to 24 hours postoperatively
  Time from arrival to the recovery unit until the patient's first activation of the patient-controlled analgesia (PCA) device, measured in minutes.
Number of Analgesic Demands | 24 hours postoperatively
  Total number of times the patient activates the patient-controlled analgesia (PCA) device to request analgesic medication during the postoperative period.
Need for Rescue Analgesia | 24 hours postoperatively
  Incidence of rescue analgesia requirement (defined as NRS pain score ≥4) and total dose of rescue analgesic medications administered outside of the PCA protocol, including medication type and dose.
Incidence and Severity of Postoperative Nausea and Vomiting (PONV) | 24 hours postoperatively
  Assessment of postoperative nausea and vomiting using the Postoperative Nausea Vomiting Impact Scale Score, evaluating both incidence and severity.
Patient Satisfaction Score | 24 hours postoperatively
  Patient satisfaction with postoperative pain management assessed on a 6-point scale (0 = not satisfied at all, 5 = very satisfied).
Time to First Mobilization | From end of surgery up to 48 hours postoperatively
  Time from the end of surgery until the patient is able to mobilize (stand and walk) for the first time, measured in hours.
Hospital Length of Stay | From surgery date until hospital discharge, assessed up to 7 days
  Duration of hospitalization from the time of surgery until hospital discharge, measured in days.
Block Efficacy Assessment | 30 minutes after ESP block administration (preoperatively)
  Dermatomal coverage and sensory block effectiveness assessed using hot-cold discrimination test at 30 minutes after block administration in the preoperative area.

CONTACTS AND LOCATIONS:
Locations (1):
- Başakşehir Çam Ve Sakura Şehir Hastanesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Koplewicz HS. From the Editor-in-Chief's Desk. J Child Adolesc Psychopharmacol. 2018 Jun;28(5):297. doi: 10.1089/cap.2018.29149.hsk. No abstract available. PMID 29889567
- [Result] Ivanusic J, Konishi Y, Barrington MJ. A Cadaveric Study Investigating the Mechanism of Action of Erector Spinae Blockade. Reg Anesth Pain Med. 2018 Aug;43(6):567-571. doi: 10.1097/AAP.0000000000000789. PMID 29746445
- [Result] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016